# Clinical Evaluation of a Manufacturing Process for a Frequent Replacement Silicone Hydrogel Multifocal Contact Lens

STUDY ID

CLN705-M103

**PROTOCOL** 

NCT05765227



# Feasibility Clinical Protocol for CLN705-M103 Title: Clinical evaluation of a manufacturing process for a frequent replacement silicone hydrogel multifocal contact lens

| Protocol Number and Version: | CLN705-M103, Version 1.0 |
|---|---|
| Sponsor Name and Address: | Alcon Research, LLC and its affiliates ("Alcon") 6201 South Freeway Fort Worth, Texas 76134-2099 |
| Test Product(s): | Lehfilcon A Multifocal SiHy contact lens |
| | Air Optix plus Hydraglyde MF contact lens (AOHG MF) |

#### **Sponsor Contact Details**



Property of Alcon
Confidential
May not be used, divulged, published, or otherwise disclosed without the consent of
Alcon

Document ID: V-CLN-0038373

Status: Approved, Version: 1.0 Page 2 of 21 Approved Date: 22 Feb 2023

Investigator Agreement:

| • | I have read the Feasibility Clinical Protocol described herein and the |
|---|---|
| | Feasibility Clinical Protocol governing it, recognize its confidentiality, and |
| | agree to conduct the described trial in compliance with Good Clinical Practice |
| | (GCP), the ethical principles contained within the Declaration of Helsinki, this |
| | protocol, all applicable regulatory authority regulations, and conditions of approval |
| | imposed by the reviewing IRB or regulatory authority. |

- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current Investigator's Brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authority? | | |
|---|---|---|---|
| | □ No □ | Yes | |
| | Have you ev | er been involved in a study or other researc | h that was terminated? |
| | □ No □ | Yes | |
| | If yes, please explain here: | | |
| Pr | incipal investi | gator: | |
| | | Signature | Date |
| | me and profesition: | ssional | |
| Αc | ldress: | | |

# **Table of Contents**

| Feasibility ( | Clinical Protocol for CLN705-M103 | 1 |
|---------------|----------------------------------------------|----|
| Table of Co | ontents | 3 |
| | les | |
| Abbreviatio | ons and Acronyms | 4 |
| 1 FEASIE | BILITY CLINICAL PROTOCOL | 5 |
| 1.1 | Revision History | 5 |
| 1.2 | Study Overview | 5 |
| 1.3 | Study Product and Associated Materials | 11 |
| 1.4 | Study-Specific Lens Returns | 19 |
| | 1.4.1 Worn IP | 19 |
| | List of Tables | |
| Table 1-1 | Schedule of Study Procedures and Assessments | 14 |

| Table 1-1 | Schedule of Study | Procedures and Assessments | l | L Z |
|-----------|-------------------|----------------------------|---|-----|
|-----------|-------------------|----------------------------|---|-----|

# **Abbreviations and Acronyms**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| °C | Degrees Celsius |
| CDMA | Clinical Development & Medical Affairs |
| CSS | Clinical Site Specialist |
| CT&OL | Clinical Trial & Operations Lead |
| D | Diopter(s) |
| eCRF | Electronic case report form |
| GA | Georgia |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| ID | Identification |
| IP | Investigational product |
| IRB | Institutional review board |
| JCR | Johns Creek Research |
| LID | Lens identification number |
| logMAR | Logarithm of the minimum angle of resolution |
| MR | Manifest refraction |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |
| PI | Principal investigator |
| R&D | Research & Development |
| SADE | Serious adverse device effect |
| SiHy | Silicone hydrogel |
| US or USA | United States |

| Abbreviation | Definition |
|--------------|---------------|
| VA | Visual acuity |

# 1 FEASIBILITY CLINICAL PROTOCOL

# 1.1 Revision History

| Version | Brief Description and Rationale |
|---------|----------------------------------|
| 1 | Initial Version of this document |

#### 1.2 Study Overview

| Protocol Study Details | | |
|---|---|---|
| Study Rationale and Objective | The purpose of this clinical trial is to evaluate the clinical performance of a manufacturing process on a frequent replacement multifocal contact lens | |
| Investigator(s) Site | Johns Creek Research Clinic<br>11460 Johns Creek Parkway<br>Johns Creek, GA, 30097 USA | |
| External Organizations | Not Applicable | |
| Planned Duration of Exposure | Subjects will be exposed to up to 2 be worn for 2 days (+3 days): • Study Lens 1 | study lenses per eye, each will |
| Number of Subjects | Planned to enroll: Up to 150 subjects Target to complete: Up to 150 subjects | |
| Study Population | <ul> <li>Habitual soft Multifocal contact lens wearers aged ≥ 40 years with normal eyes (not needing ocular medication, other than correction for refractive error). Subjects should have at least 3 months wearing experience, wear these lenses at least 5 days per week and at least 8 hours per day.</li> <li>To qualify, subjects must require cylindrical correction ≤ 0.75D, be able wear study contact lens with sphere power ranging</li> </ul> | |

| Ducto cal Study Dataila | | |
|---|---|---|
| Protocol Study | | |
| | | and requiring a near ADD of LO, |
| • | MED or HI | |
| Lens Assignment | No formal randomization will be | implemented (a predetermined |
| | order will be provided by Sponso | |
| Study Design | Prospective | Single-masked (trial subject) |
| Study Design | | |
| | Randomized | Open-label |
| | Single group | Contralateral |
| | Parallel group | |
| | Crossover | Monocular lens wear |
| | Other: either single group or | |
| | crossover depending on number | |
| | of study lenses evaluated | |
| | Visit Schedule: | |
| | • If only 1 study lens to be tested in a trial: | |
| | 1. Visit 1 - Screening/Baseline/Dispense Lens 1 | |
| | 2. Visit 2 (2 (+3) days after Visit 1) Follow-up Lens 1 (to occur at least 4-6 hours after lens insertion)/Exit | |
| | occur at least 4-6 hours after lens hisertion)/Exit | |
| <b>Decision Criteria</b> | No prospective decision criteria have been defined for this study. | |
| Assessments | 1. VA with study lenses (logMAR; OU) @ 4m | |



| Protocol Study Details | |
|---|---|
| | 6. BCVA 0.1 logMAR or better in each eye. |
| | 7. Able to fit with available contact lenses: within a range of powers from +3.00D to -7.00 and requiring a near ADD of LO, MED or HI, as available |
| | 8. Subject must possess spectacles that provide a corrected visual acuity of 20/40 or better OU. |
| Exclusion Criteria | 1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator. |
| | 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator. |
| | 3. History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye. |
| | 4. Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study. |
| | 5. Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher, and/or any infiltrate. |
| | 6. Current or history of pathologically dry eye in either eye that, in the opinion of the investigator, would preclude contact lens wear. |
| | 7. Current or history of herpetic keratitis in either eye. |
| | 8. Eye injury in either eye within 12 weeks immediately prior to enrollment for this trial. |
| | 9. Current or history of intolerance, hypersensitivity, or allergy to any component of the study products. |
| | 10. The investigator, his/her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of the aforementioned persons in the study. |
| | 11. Participation of the subject in a clinical trial within the previous 2 days or currently enrolled in any clinical trial. |
| | 12. Monovision contact lens wearer |
| Enrollment<br>Stopping Criteria | Enrollment stopping criteria will not be defined for this study. |
| | Analysis Plan |
| Statistical Analysis | |

| Protocol Study Details | | | |
|---|---|---|---|
| | The following product or lens naming conventions will be used: AOHG MF | | |
| Subject Characteristics and Study Conduct Summaries | The following will be presented: • Conduct | | |
| Assessment<br>Analysis Strategy | Results from selected assessment will be summarized using descriptive statistics according to its measurement scale. Listings will be provided as necessary. The Safety Analysis Set will serve as the analysis data set for all effectiveness analyses. | | |
| Planned<br>Effectiveness<br>Analyses | Title VA with study lenses | Assessment Visual Acuity • 4m (OU) | Analysis Table for continuous variables (Dispense, Follow-up) |

| Protocol Study Details | |
|---|---|
| Sample Size and Power | No formal sample size calculation is provided given the descriptive and feasibility nature of the study. |
| Calculations | and reasionity nature of the study. |

# 1.3 Study Product and Associated Materials

| | Test Product 1 MF contact lenses or LID | Comparator Product 1<br>[AIR OPTIX plus<br>HydraGlyde Multifocal] |
|---|---|---|
| Primary<br>component/<br>material | Lehfilcon A | Lotrafilcon B |
| Manufacturer | Alcon Laboratories, Inc. | Alcon Laboratories, Inc. |
| Power Range | <ul> <li>LO Add with +1.00 to -5.00D (in 0.25D steps) spherical power as available</li> <li>MED Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> <li>HI Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> </ul> | <ul> <li>LO Add with +1.00 to -5.00D (in 0.25D steps) spherical power as available</li> <li>MED Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> <li>HI Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> </ul> |
| Supply | The sponsor will provide this test product. | The site will procure this comparator product. |
| Packaging and<br>Labeling | Primary label on blister foil pack includes, at a minimum: • material name or identifier • base curve | Commercial primary and secondary labeling and packaging |

| | Test Product 1 MF contact lenses or LID | Comparator Product 1 [AIR OPTIX plus HydraGlyde Multifocal] |
|---|---|---|
| | include the following] Commercial primary label on blister foil pack includes: • material name • base curve • diameter • packing solution • power • lot number • expiration date • content statement • country of origin • manufacturer information | |
| Storage | Lenses should be stored at room temperature. | Refer to manufacturer's instructions. |
| Other | Replacement lenses are allowed only if there is a device deficiency (e.g., torn lens) or if the lens falls on the ground and investigator wants to insert a new lens. | Replacement lenses are allowed only if there is a device deficiency (e.g., torn lens) or if the lens falls on the ground and investigator wants to insert a new lens. |
| Associated | CLEAR CARE Cleaning | g and Disinfecting Solution will be used with study |

| Status: Approved, Version: 1.0 |
|--------------------------------|
| Approved Date: 22 Feb 2023 |

| | Test Product 1 MF contact lenses or LID | Comparator Product 1 [AIR OPTIX plus HydraGlyde Multifocal] |
|---|---|---|
| Materials | lenses for the duration of study. | |
| | • LacriPure rinsing/reinsertion PRN will be used as needed with study lenses. | |
| | • Lubrication/re-wetting drops will not be permitted during study lens wear. | |

 Table 1-1
 Schedule of Study Procedures and Assessments

| | | Visit 1 | Visi | t 2 | | | |
|---|---|---|---|---|---|---|---|
| | Procedure/ Assessment | Screening/Baseline/<br>Dispense Lens 1 | Follow up Lens 1 (2 (+ 3) Days) after Visit 1 (minimum 4 - 6 hrs after insertion) | | Exit | Unscheduled<br>Visit/Early<br>Exit Visit | Source<br>Only* |
| 1 | Informed Consent | X | | | | | |
| 2 | Demographics | X | | | | | |
| 3 | Medical History | X | X | | | X | X |
| 4 | <b>Concomitant Medications</b> | X | X | | | X | X |
| 5 | Inclusion/ Exclusion | X | | | | | |
| 6 | Habitual lens (brand, power) | X | | | | | |
| 7 | VA w/ habitual correction (OD, OS, Snellen distance) | X | (X) | | X | (X) | X |
| 8 | Manifest refraction (most plus sphero-<br>cylindrical)<br>(data for repeat subjects – ILB in EDC) | X | | | (X) | (X) | |
| 9 | BCVA (OD, OS, logMAR; distance and near with manifest refraction) | X | | | (X) | (X) | |
| 10 | Biomicroscopy | X | X | | | X | |

| 1 | | | | | | |
|---|---|---|---|---|---|---|
| | | Visit 1 | Visit 2 | | Unscheduled | |
| | Procedure/ Assessment | Screening/Baseline/<br>Dispense Lens 1 | Follow up Lens 1<br>(2 (+ 3) Days) after<br>Visit 1<br>(minimum 4 - 6 hrs<br>after insertion) | Exit | Visit/Early<br>Exit Visit | Source<br>Only* |
| 13 | Dispense study lenses | X | | | (X) | X |
| 17 | VA w/ study lenses, (logMAR) • Distance (4m; OU) | X | X | | (X) | |

Page 17 of 21

Visit 2 Visit 1 Unscheduled Source Follow up Lens 1 Exit Visit/Early **Procedure/ Assessment** Only\* (2 (+ 3) Days) after Visit 1 Screening/Baseline/ **Exit Visit** Dispense Lens 1 (minimum 4 - 6 hrs after insertion) **Collect worn lenses** X (X) 28 **AEs** X X X X X X X X **Device deficiencies** 

Status: Approved, Version: 1.0

Approved Date: 22 Feb 2023

| | Procedure/ Assessment | Visit 1 | Visi | t 2 | | Unscheduled | |
|---|---|---|---|---|---|---|---|
| | | Screening/Baseline/<br>Dispense Lens 1 | Follow up Lens 1<br>(2 (+ 3) Days) after<br>Visit 1<br>(minimum 4 - 6 hrs<br>after insertion) | | Exit | Visit/Early Exit Visit | Source<br>Only* |
| 30 | Exit Form | (X) | (X) | | X | (X) | |

#### 1.4 Study-Specific Lens Returns

#### 1.4.1 Worn IP

Worn IP will be returned to the sponsor. Use the following instructions for collection, storage, and shipping, unless otherwise instructed by the sponsor.

If worn IP is to be returned, provide all of the following specifications:

- Removal from eye: Clean hands
- Storage container: Unused screw-top lens case
- Label information:
  - Protocol number
  - o Site number
  - Subject ID
  - o Eye
  - Lens type/ identification
  - Lot number
  - o Date collected
- Storage solution: PURILENS Plus Preservative Free Saline (PURILENS Plus Saline)
- Storage temperature: Refrigerated 4-10°C
- Timing of return: Study Completion or periodically as communicated by sponsor
- An inventory/list of lenses being returned



